CLINICAL TRIAL: NCT00710840
Title: Functional Outcomes Following Minimally Invasive Total Knee Arthroplasty
Brief Title: Effectiveness of Minimally Invasive Total Knee Replacement in Improving Rehabilitation and Function
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-0183; R03AR054538 (NIH); 1R03AR054538-01A2 (NIH)
Record Dates: First submitted 2008-06-27; First posted 2008-07-04 (Estimated); Results first posted 2015-05-15 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-03

CONDITIONS: Osteoarthritis
Keywords: Knee Replacement; Knee OA; OA
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroplasty, Replacement, Knee

ARMS (2):
- 1 (Experimental)
  Interventions: Procedure: Minimally Invasive Total Knee Arthroplasty [TKA Min]
- 2 (Active Comparator)
  Interventions: Procedure: Total Knee Arthroplasty (TKA) Traditional

INTERVENTIONS:
Procedure: Minimally Invasive Total Knee Arthroplasty [TKA Min] — TKA Min is a procedure in which diseased and painful joint surfaces of the knee are replaced by metal and plastic components shaped to allow continued motion of the knee. TKA Min, as opposed to TKA Traditional, employs smaller skin incisions and smaller instrumentation and avoids turning the knee cap out and dislocating the knee. This procedure also avoids disrupting the knee extensor mechanism and the suprapatellar pouch and minimizes extreme knee flexion during surgery.
  Other Names: TKA Min
  Arms: 1
Procedure: Total Knee Arthroplasty (TKA) Traditional — TKA is a procedure in which diseased and painful joint surfaces of the knee are replaced by metal and plastic components shaped to allow continued motion of the knee.
  Other Names: TKA Traditional
  Arms: 2

SUMMARY:
Osteoarthritis (OA) is a long-term degenerative joint disease that disables about 10% of people over the age of 60 and compromises the quality of life of more than 20 million Americans. A procedure called total knee arthroplasty (TKA), in which the affected surface of the knee joint is replaced by plastic or metal, has been successful in restoring comfort and mobility to formerly arthritic joints. This study will compare quadriceps muscle strength, knee range of motion, and pain in people who have had a traditional TKA with those who have had a minimally invasive TKA.

DETAILED DESCRIPTION:
More than 400,000 TKAs are performed each year in the United States to alleviate pain and disability associated with knee OA. Although this procedure reliably reduces pain and improves function in people with knee OA, recovery of the strength of the quadriceps muscle to normal levels is rare. For years after a TKA, performance while walking or while doing a more physically demanding activity, such as stair climbing, is also significantly lower in people who have had a TKA than in healthy adults of the same age. Within the past few years, less invasive TKA surgical techniques have been developed as promising alternatives to traditional TKA. Minimally invasive TKA, or TKA(min), achieves the same surgical objectives, but possibly without doing as much damage to the quadriceps muscle as is seen with traditional TKA. No studies, however, have specifically investigated how TKA(min) might preserve quadriceps muscle function. This study will determine whether TKA(min) is better than TKA at improving quadriceps muscle force production and activation, increasing knee range of motion, and reducing post-operative pain to improve overall functional outcomes.

Participants who are scheduled to undergo knee replacement surgery will be randomly assigned to receive either traditional TKA or TKA(min). Prior to surgery, participants will attend a 30-minute orientation session and undergo certain tests to evaluate knee function. Functional testing will include timed walking, stair climbing, balance testing, and knee flexibility measurements. Other evaluations will include thigh muscle strength and activation testing, which uses brief electrical pulses to determine if the muscles are contracted as much as possible, and health status questionnaires. After the operation, participants will be instructed to use walking aids, such as a walker, crutches, or a cane, for a period of time. Participants will attend study visits for repeat testing 48 hours following surgery; at Months 1, 3, and 6; and at Years 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of osteoarthritis
* Eligible for a unilateral or bilateral primary TKA to be performed by Dr. Michael Dayton (University of Colorado Hospital)
* Minimum of 110 degrees of active knee flexion
* No greater than 10 degrees of anatomic knee varus, 15 degrees anatomic valgus, and 10 degrees flexion contracture
* Body mass index less ≤ 40 kg/m2

Exclusion Criteria:

* Any brain, circulation, or heart problems that limit function
* Severe osteoarthritis or other orthopedic conditions that limit function in the lower extremity that is not undergoing the TKA

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-06; Primary Completion 2011-02 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer E. Stevens, MPT, PhD, Principal Investigator — University of Colorado, Denver; Michael Dayton, MD, Principal Investigator — University of Colorado, Denver; Wendy Kohrt, PhD, Principal Investigator — University of Colorado School of Medicine
Locations (3):
- United States (3):
  - University of Colorado Health Sciences Center, Boulder, Colorado
  - National Jewish Medical and Research Center, Denver, Colorado
  - University of Colorado Health Sciences Center, Denver, Colorado

RESULTS

PARTICIPANT FLOW:
Groups:
- TKA Min: Minimally Invasive Total Knee Arthroplasty [TKA(min)]: TKA(min) is a procedure in which diseased and painful joint surfaces of the knee are replaced by metal and plastic components shaped to allow continued motion of the knee. TKA(min), as opposed to TKA, employs smaller skin incisions and smaller instrumentation and avoids turning the knee cap out and dislocating the knee. This procedure also avoids disrupting the knee extensor mechanism and the suprapatellar pouch and minimizes extreme knee flexion during surgery.
- TKA Traditional: Total Knee Arthroplasty (TKA): TKA is a procedure in which diseased and painful joint surfaces of the knee are replaced by metal and plastic components shaped to allow continued motion of the knee.
Period: Overall Study
Arm/Group | TKA Min | TKA Traditional
Started | 22 | 22
Completed | 22 | 19
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TKA Min | TKA Traditional | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (8.5) | 64.0 (8.4) | 64.3 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 10 | 12 | 22
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 44
BMI [Mean (Standard Deviation); unit: kg\m^2] | 30.5 (5.6) | 31.3 (5.1) | 30.9 (5.4)

OUTCOME MEASURES:

1. Primary Outcome: Quadriceps Muscle Force
Time Frame: Measured pre-operatively; post-surgery at 4 weeks and 12 weeks
Measure: Mean (Standard Deviation); unit: Nm/kg
Arm/Group | TKA Min | TKA Traditional
Number analyzed (Participants) | 22 | 19
Nm/kg
  Quadriceps Strength Preop | 1.27 (0.56) | 1.37 (0.56)
  Quadriceps Strength 4 weeks Postop | 0.79 (0.39) | 0.66 (0.23)
  Quadriceps Strength 12 weeks Postop | 1.24 (0.40) | 1.20 (0.42)
Statistical Analysis 1: Comparison: TKA Min vs TKA Traditional; The primary outcome, difference in quadriceps torque between intervention (TKA Min) and Control TKA at 4 weeks, was tested using an analysis of covariance model. Confirmatory measures were evaluated at 4 and 12 weeks after surgery in the same way. Baseline characteristics of the treatment groups were compared using 2-sample t tests for continuous measures or a χ2 test for independent proportions for categorical measures. A 2-sided α level of .05 was designated for statistical significance; Test type: Superiority or Other; p = 0.07, t-test, 2 sided — Difference in the change from Preop to 4 weeks Postop

2. Secondary Outcome: Functional Performance: 6 Minute Walk (6MW) Distance
Time Frame: Measured pre-operatively; post-surgery at 4 weeks and 12 weeks
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | TKA Min | TKA Traditional
Number analyzed (Participants) | 22 | 19
Meters
  6MW Preop | 464.0 (124.9) | 434.7 (147.8)
  6MW 4 weeks Postop | 345.9 (111.2) | 326.6 (125.7)
  6MW 12 weeks Postop | 474.6 (105.4) | 448.5 (124.8)
Statistical Analysis 1: Comparison: TKA Min vs TKA Traditional; Test type: Superiority or Other; p = 0.92, t-test, 2 sided — Difference in the change from Preop to 4 weeks Postop

3. Primary Outcome: Knee Range of Motion
Description: Knee Flexion Active Range of Motion (AROM)
Time Frame: Measured pre-operatively; post-surgery at 4 weeks and 12 weeks
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | TKA Min | TKA Traditional
Number analyzed (Participants) | 22 | 19
degrees
  Flexion AROM Preop | 120.0 (16.7) | 119.3 (15.8)
  Flexion AROM 4 weeks Postop | 98.6 (12.3) | 96.9 (13.9)
  Flexion AROM 12 weeks Postop | 113.5 (10.6) | 112.4 (9.4)
Statistical Analysis 1: Comparison: TKA Min vs TKA Traditional; Test type: Superiority or Other; p = 0.48, t-test, 2 sided — Difference in the change from Preop to 4 weeks Postop

4. Secondary Outcome: Functional Performance: Stair Climb Test
Description: This outcome measures the time (seconds) it takes to climb up and back down 12 steps.
Time Frame: Measured pre-operatively; post-surgery at 4 weeks and 12 weeks
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | TKA Min | TKA Traditional
Number analyzed (Participants) | 22 | 19
Seconds
  Stair Climb Preop | 18.1 (9.7) | 19.4 (17.2)
  Stair Climb 4 weeks Postop | 35.0 (18.7) | 32.2 (17.3)
  Stair Climb 12 weeks Postop | 15.9 (8.7) | 16.4 (7.8)
Statistical Analysis 1: Comparison: TKA Min vs TKA Traditional; Test type: Superiority or Other; p = 0.41, t-test, 2 sided — Difference in the change from Preop to 4 weeks Postop

ADVERSE EVENTS:
Arm/Group | TKA Min | TKA Traditional
Serious Adverse Events (participants affected / at risk) | 1/22 | 0/22
Other Adverse Events (participants affected / at risk) | 10/22 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TKA Min (N=22) | TKA Traditional (N=22)
Pulmonary Embolus (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TKA Min (N=22) | TKA Traditional (N=22)
Femoral Notching (Surgical and medical procedures) | 2 | 2
Retained Cement (Surgical and medical procedures) | 1 | 2
Heterotopic Ossification (Surgical and medical procedures) | 0 | 1
Retained Drill Bit (Surgical and medical procedures) | 0 | 1
Intra-Operative Fracture (Surgical and medical procedures) | 0 | 1 — Medial Condyle Fracture
Hematoma\Excessive Bleeding (Blood and lymphatic system disorders) | 2 | 6
Cellulitis (Skin and subcutaneous tissue disorders) | 0 | 2
Poor Bone Quality (General disorders) | 0 | 1 — Prevented full weight bearing after surgery
Urinary Tract Infection (Infections and infestations) | 0 | 1 — Post-op
Transient EKG Abnormality (Cardiac disorders) | 0 | 1 — Post-op
Hypersensitivity to Light Touch (Nervous system disorders) | 1 | 0
Surgical Malalignment (Surgical and medical procedures) | 4 | 4 — Greater than 4 degrees of varus post-op

LIMITATIONS AND CAVEATS:
Small sample size; Relatively short follow-up time

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes